CLINICAL TRIAL: NCT02512328
Title: First Experiences With an Offline App (SPA; Smartphone Application) for Colonoscopy Preparation- PERICLES-I APP; Prospective Evaluations of Improvement of Colonocopy Preparation by Optimized Visualization (PERICLES)
Brief Title: Improvement of Colonoscopy Preparation by New Media (APP)
Acronym: PERICLESAPPI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Monther Bajbouj, Physician, Technical University of Munich
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PERICLES-I-APP
Record Dates: First submitted 2015-02-24; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Colonoscopy; new media; APP; colonoscopy preparation; SPA; smartphone application
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular colonoscopy preparation (No Intervention): Comparison group. Regular colonoscopy preparation
- APP supported colonoscopy preparation (Experimental): APP as additional device for colonoscopy preparation
  Interventions: Device: APP supported colonoscopy preparation

INTERVENTIONS:
Device: APP supported colonoscopy preparation — additional usage of an app for colonoscopy preparation
  Arms: APP supported colonoscopy preparation

SUMMARY:
Feasibility of an newly programmed offline application for smartphones (SPA, APP) for colonoscopy preparation offering a 5 day guidance prior colonoscopy containing dietary- and behavioral recommendation.

DETAILED DESCRIPTION:
First feasibility testing of a newly programmed app/SPA for android system named Colopr-APP. It is an strictly offline working, autonomous system downloaded to the smartphone. It creates an 5-day guidance prior outpatient colonoscopy with dietary and behavior recommendations.

ELIGIBILITY:
Inclusion Criteria:

* outpatient colonoscopy
* smartphone owner with android system

Exclusion Criteria:

* chronic renal failure
* anticoagulants
* pregnancy
* diabetes mellitus (IDDM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility | at day 0 colonoscopy after colonoscopy preparation
  feasibility of app supported colonoscopy preparation (stable working and function of software on smartphone)

SECONDARY OUTCOMES:
Bowel preparation | at day 0 after colonoscopy
  Evaluation of bowel preparation during colonoscopy by BostenBowelPreparation Scale
patient´s satification | day 1 after colonoscopy
  Evaluation of patient´s satisfication by a questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Walter, MD, Principal Investigator — Physician
Locations (1):
- 2nd Medical Department, Klinikum rechts der Isar, Munich, Germany

REFERENCES:
- [Derived] Walter B, Schmid R, von Delius S. A Smartphone App for Improvement of Colonoscopy Preparation (ColoprAPP): Development and Feasibility Study. JMIR Mhealth Uhealth. 2017 Sep 20;5(9):e138. doi: 10.2196/mhealth.7703. PMID 28931498